CLINICAL TRIAL: NCT02058927
Title: Immune Reconstitution to Measles Virus of HIV-1-Infected Zambian Children Initiating Antiretroviral Therapy
Brief Title: Immune Reconstitution to Measles Virus of HIV Infected Children in Zambia
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Carolyn Bolton Moore, MD, Assistant Professor, University of North Carolina, Chapel Hill
Other Study IDs: CIDRZ 1204/IRB12-0400; R01AI070018 (NIH)
Record Dates: First submitted 2014-02-06; First posted 2014-02-10 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Measles
Keywords: HIV; ART; children
MeSH Terms: conditions — Measles | interventions — Measles Vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples will be stored in a repository for five years beyond the end of the study period. Some samples may be exported to the Johns Hopkins Bloomberg School of Public Health when assays cannot be performed in Zambia.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- HIV-1 infected children: HIV-1-infected children initiating ART
- HIV-1 uninfected children: control group of HIV-1 uninfected children matched by age
- HIV-1 infected children revaccinated: nested study of revaccination against measles virus of HIV-1-infected children receiving ART who lack protective antibody titers
  Interventions: Drug: Measles vaccine

INTERVENTIONS:
Drug: Measles vaccine — measles revaccination administered at 12 months from start of ART
  Groups: HIV-1 infected children revaccinated

SUMMARY:
This is an observational study of HIV-1 infected children starting antiretroviral therapy to measure the magnitude and quality of general immune reconstitution and pathogen-specific immune reconstitution to measles virus.

DETAILED DESCRIPTION:
This is a prospective, observational cohort study of 230 HIV-1-infected children initiating ART at public clinics in Lusaka, Zambia to measure the magnitude and quality of general immune reconstitution and pathogen-specific immune reconstitution to measles virus. Non-specific immune reconstitution will be assessed by serial measurements of the number and percentages of CD4+ and CD8+ T-lymphocytes, number and percentages of activated CD4+ and CD8+ T-lymphocytes (using cell surface staining for HLA-DR and CD38), changes in the proportions of naïve and memory CD4+ and CD8+ T-lymphocyte subsets (using cell surface staining for CD45RA and CCR7), and changes in thymic output as determined by TREC levels. Virologic responses to ART will be assessed by serial measurements of plasma HIV-1 RNA levels.

Within the observational study, there is a nested study of revaccination against measles virus of HIV-1-infected children receiving ART who lack protective antibody titers to assess the proportion of revaccinated children who develop protective immunity and the duration of protective immunity. Anti-measles virus IgG antibodies will be measured 9 months after initiation of ART. The results will be available at the 12-month follow-up visit and measles revaccination will be recommended to those children lacking protective antibody levels to measles virus.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls 9 months to 10 years of age residing in Lusaka, Zambia are eligible for enrolment.
* initiating ART
* history of measles vaccination confirmed by examination of the Immunization Card.

Ages: 9 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: HIV-1 infected children initiating ART in public clinics within Lusaka, Zambia.
Sampling Method: Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2011-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Memory immune responses to measles virus | 0, 6, 12, 24, 30 and 36 months from start of ART
  Memory immune responses to measles virus will be measured to characterize the magnitude and quality of immune reconstitution in HIV-1 infected Zambian children initiating ART and determine pathogen-specific immune reconstitution.

SECONDARY OUTCOMES:
Humoral and cellular immune responses to measles virus before and after revaccination | 12, 15, 24, 30 and 36 months from start of ART
  Humoral and cellular immune responses to measles virus before and after revaccination of HIV-1-infected Zambian children receiving ART who lack protective antibody titers will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn B Moore, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Centre for Infectious Disease Research in Zambia, Lusaka, Zambia

REFERENCES:
- [Background] Newell ML, Brahmbhatt H, Ghys PD. Child mortality and HIV infection in Africa: a review. AIDS. 2004 Jun;18 Suppl 2:S27-34. doi: 10.1097/00002030-200406002-00004. PMID 15319741
- [Background] de Martino M, Tovo PA, Balducci M, Galli L, Gabiano C, Rezza G, Pezzotti P. Reduction in mortality with availability of antiretroviral therapy for children with perinatal HIV-1 infection. Italian Register for HIV Infection in Children and the Italian National AIDS Registry. JAMA. 2000 Jul 12;284(2):190-7. doi: 10.1001/jama.284.2.190. PMID 10889592
- [Background] Gortmaker SL, Hughes M, Cervia J, Brady M, Johnson GM, Seage GR 3rd, Song LY, Dankner WM, Oleske JM; Pediatric AIDS Clinical Trials Group Protocol 219 Team. Effect of combination therapy including protease inhibitors on mortality among children and adolescents infected with HIV-1. N Engl J Med. 2001 Nov 22;345(21):1522-8. doi: 10.1056/NEJMoa011157. PMID 11794218
- [Background] Autran B, Carcelain G, Li TS, Blanc C, Mathez D, Tubiana R, Katlama C, Debre P, Leibowitch J. Positive effects of combined antiretroviral therapy on CD4+ T cell homeostasis and function in advanced HIV disease. Science. 1997 Jul 4;277(5322):112-6. doi: 10.1126/science.277.5322.112. PMID 9204894
- [Background] Pakker NG, Notermans DW, de Boer RJ, Roos MT, de Wolf F, Hill A, Leonard JM, Danner SA, Miedema F, Schellekens PT. Biphasic kinetics of peripheral blood T cells after triple combination therapy in HIV-1 infection: a composite of redistribution and proliferation. Nat Med. 1998 Feb;4(2):208-14. doi: 10.1038/nm0298-208. PMID 9461195
- [Background] Gibb DM, Newberry A, Klein N, de Rossi A, Grosch-Woerner I, Babiker A. Immune repopulation after HAART in previously untreated HIV-1-infected children. Paediatric European Network for Treatment of AIDS (PENTA) Steering Committee. Lancet. 2000 Apr 15;355(9212):1331-2. doi: 10.1016/s0140-6736(00)02117-6. PMID 10776748
- [Background] Vigano A, Vella S, Saresella M, Vanzulli A, Bricalli D, Di Fabio S, Ferrante P, Andreotti M, Pirillo M, Dally LG, Clerici M, Principi N. Early immune reconstitution after potent antiretroviral therapy in HIV-infected children correlates with the increase in thymus volume. AIDS. 2000 Feb 18;14(3):251-61. doi: 10.1097/00002030-200002180-00007. PMID 10716501
- [Background] van Rossum AM, Scherpbier HJ, van Lochem EG, Pakker NG, Slieker WA, Wolthers KC, Roos MT, Kuijpers JH, Hooijkaas H, Hartwig NG, Geelen SP, Wolfs TF, Lange JM, Miedema F, de Groot R; Dutch Study Group for Children with HIV Infections. Therapeutic immune reconstitution in HIV-1-infected children is independent of their age and pretreatment immune status. AIDS. 2001 Nov 23;15(17):2267-75. doi: 10.1097/00002030-200111230-00008. PMID 11698700
- [Background] Douek DC, Koup RA, McFarland RD, Sullivan JL, Luzuriaga K. Effect of HIV on thymic function before and after antiretroviral therapy in children. J Infect Dis. 2000 Apr;181(4):1479-82. doi: 10.1086/315398. Epub 2000 Apr 13. PMID 10762580
- [Background] Chavan S, Bennuri B, Kharbanda M, Chandrasekaran A, Bakshi S, Pahwa S. Evaluation of T cell receptor gene rearrangement excision circles after antiretroviral therapy in children infected with human immunodeficiency virus. J Infect Dis. 2001 May 15;183(10):1445-54. doi: 10.1086/320197. Epub 2001 Apr 13. PMID 11329124
- [Background] Johnston AM, Valentine ME, Ottinger J, Baydo R, Gryszowka V, Vavro C, Weinhold K, St Clair M, McKinney RE. Immune reconstitution in human immunodeficiency virus-infected children receiving highly active antiretroviral therapy: a cohort study. Pediatr Infect Dis J. 2001 Oct;20(10):941-6. doi: 10.1097/00006454-200110000-00006. PMID 11642627
- [Background] De Rossi A, Walker AS, Klein N, De Forni D, King D, Gibb DM. Increased thymic output after initiation of antiretroviral therapy in human immunodeficiency virus type 1-infected children in the Paediatric European Network for Treatment of AIDS (PENTA) 5 Trial. J Infect Dis. 2002 Aug 1;186(3):312-20. doi: 10.1086/341657. Epub 2002 Jul 5. PMID 12134227
- [Background] Resino S, Correa R, Bellon JM, Sanchez-Ramon S, Munoz-Fernandez MA. Characterizing immune reconstitution after long-term highly active antiretroviral therapy in pediatric AIDS. AIDS Res Hum Retroviruses. 2002 Dec 10;18(18):1395-406. doi: 10.1089/088922202320935474. PMID 12487811
- [Background] Burgess K, Price P, James IR, Stone SF, Keane NM, Lim AY, Warmington JR, French MA. Interferon-gamma responses to Candida recover slowly or remain low in immunodeficient HIV patients responding to ART. J Clin Immunol. 2006 Mar;26(2):160-7. doi: 10.1007/s10875-006-9008-4. Epub 2006 Mar 28. PMID 16568352
- [Background] Hainaut M, Ducarme M, Schandene L, Peltier CA, Marissens D, Zissis G, Mascart F, Levy J. Age-related immune reconstitution during highly active antiretroviral therapy in human immunodeficiency virus type 1-infected children. Pediatr Infect Dis J. 2003 Jan;22(1):62-9. doi: 10.1097/00006454-200301000-00016. PMID 12544411
- [Background] Weinberg A, Pahwa S, Oyomopito R, Carey VJ, Zimmer B, Mofenson L, Kovacs A, Burchett SK; Pediatric AIDS Clinical Trials Group 366 Team. Antimicrobial-specific cell-mediated immune reconstitution in children with advanced human immunodeficiency virus infection receiving highly active antiretroviral therapy. Clin Infect Dis. 2004 Jul 1;39(1):107-14. doi: 10.1086/420931. Epub 2004 Jun 14. PMID 15206061
- [Background] Weinberg A, Wiznia AA, LaFleur BJ, Shah S, Levin MJ. Varicella-Zoster virus-specific cell-mediated immunity in HIV-infected children receiving highly active antiretroviral therapy. J Infect Dis. 2004 Jul 15;190(2):267-70. doi: 10.1086/422011. Epub 2004 Jun 9. PMID 15216460
- [Background] Weinberg A, Gona P, Nachman SA, Defechereux P, Yogev R, Hughes W, Wara D, Spector SA, Read J, Elgie C, Cooper M, Dankner W; Pediatric AIDS Clinical Trials Group 1008 Team. Antibody responses to hepatitis A virus vaccine in HIV-infected children with evidence of immunologic reconstitution while receiving highly active antiretroviral therapy. J Infect Dis. 2006 Jan 15;193(2):302-11. doi: 10.1086/498979. Epub 2005 Dec 7. PMID 16362896
- [Background] Crotty S, Ahmed R. Immunological memory in humans. Semin Immunol. 2004 Jun;16(3):197-203. doi: 10.1016/j.smim.2004.02.008. PMID 15130504
- [Background] Lanzavecchia A, Sallusto F. Understanding the generation and function of memory T cell subsets. Curr Opin Immunol. 2005 Jun;17(3):326-32. doi: 10.1016/j.coi.2005.04.010. PMID 15886125
- [Background] Sun JC, Bevan MJ. Defective CD8 T cell memory following acute infection without CD4 T cell help. Science. 2003 Apr 11;300(5617):339-42. doi: 10.1126/science.1083317. PMID 12690202
- [Background] Shedlock DJ, Shen H. Requirement for CD4 T cell help in generating functional CD8 T cell memory. Science. 2003 Apr 11;300(5617):337-9. doi: 10.1126/science.1082305. PMID 12690201
- [Background] Janssen EM, Lemmens EE, Wolfe T, Christen U, von Herrath MG, Schoenberger SP. CD4+ T cells are required for secondary expansion and memory in CD8+ T lymphocytes. Nature. 2003 Feb 20;421(6925):852-6. doi: 10.1038/nature01441. Epub 2003 Feb 9. PMID 12594515
- [Background] Castellino F, Huang AY, Altan-Bonnet G, Stoll S, Scheinecker C, Germain RN. Chemokines enhance immunity by guiding naive CD8+ T cells to sites of CD4+ T cell-dendritic cell interaction. Nature. 2006 Apr 13;440(7086):890-5. doi: 10.1038/nature04651. PMID 16612374
- [Background] Sun JC, Williams MA, Bevan MJ. CD4+ T cells are required for the maintenance, not programming, of memory CD8+ T cells after acute infection. Nat Immunol. 2004 Sep;5(9):927-33. doi: 10.1038/ni1105. Epub 2004 Aug 8. PMID 15300249
- [Background] Kaech SM, Tan JT, Wherry EJ, Konieczny BT, Surh CD, Ahmed R. Selective expression of the interleukin 7 receptor identifies effector CD8 T cells that give rise to long-lived memory cells. Nat Immunol. 2003 Dec;4(12):1191-8. doi: 10.1038/ni1009. Epub 2003 Nov 16. PMID 14625547
- [Background] Madakamutil LT, Christen U, Lena CJ, Wang-Zhu Y, Attinger A, Sundarrajan M, Ellmeier W, von Herrath MG, Jensen P, Littman DR, Cheroutre H. CD8alphaalpha-mediated survival and differentiation of CD8 memory T cell precursors. Science. 2004 Apr 23;304(5670):590-3. doi: 10.1126/science.1092316. PMID 15105501
- [Background] McHeyzer-Williams LJ, McHeyzer-Williams MG. Antigen-specific memory B cell development. Annu Rev Immunol. 2005;23:487-513. doi: 10.1146/annurev.immunol.23.021704.115732. PMID 15771579
- [Background] Crotty S, Kersh EN, Cannons J, Schwartzberg PL, Ahmed R. SAP is required for generating long-term humoral immunity. Nature. 2003 Jan 16;421(6920):282-7. doi: 10.1038/nature01318. PMID 12529646
- [Background] Vieira P, Rajewsky K. Persistence of memory B cells in mice deprived of T cell help. Int Immunol. 1990;2(6):487-94. doi: 10.1093/intimm/2.6.487. PMID 2150759
- [Background] Hebeis BJ, Klenovsek K, Rohwer P, Ritter U, Schneider A, Mach M, Winkler TH. Activation of virus-specific memory B cells in the absence of T cell help. J Exp Med. 2004 Feb 16;199(4):593-602. doi: 10.1084/jem.20030091. Epub 2004 Feb 9. PMID 14769849
- [Background] Bernasconi NL, Traggiai E, Lanzavecchia A. Maintenance of serological memory by polyclonal activation of human memory B cells. Science. 2002 Dec 13;298(5601):2199-202. doi: 10.1126/science.1076071. PMID 12481138
- [Background] De Milito A, Morch C, Sonnerborg A, Chiodi F. Loss of memory (CD27) B lymphocytes in HIV-1 infection. AIDS. 2001 May 25;15(8):957-64. doi: 10.1097/00002030-200105250-00003. PMID 11399977
- [Background] De Milito A, Nilsson A, Titanji K, Thorstensson R, Reizenstein E, Narita M, Grutzmeier S, Sonnerborg A, Chiodi F. Mechanisms of hypergammaglobulinemia and impaired antigen-specific humoral immunity in HIV-1 infection. Blood. 2004 Mar 15;103(6):2180-6. doi: 10.1182/blood-2003-07-2375. Epub 2003 Nov 6. PMID 14604962
- [Background] Slifka MK. Immunological memory to viral infection. Curr Opin Immunol. 2004 Aug;16(4):443-50. doi: 10.1016/j.coi.2004.05.013. PMID 15245737
- [Background] Malaspina A, Moir S, Orsega SM, Vasquez J, Miller NJ, Donoghue ET, Kottilil S, Gezmu M, Follmann D, Vodeiko GM, Levandowski RA, Mican JM, Fauci AS. Compromised B cell responses to influenza vaccination in HIV-infected individuals. J Infect Dis. 2005 May 1;191(9):1442-50. doi: 10.1086/429298. Epub 2005 Mar 24. PMID 15809902
- [Background] Ovsyannikova IG, Dhiman N, Jacobson RM, Vierkant RA, Poland GA. Frequency of measles virus-specific CD4+ and CD8+ T cells in subjects seronegative or highly seropositive for measles vaccine. Clin Diagn Lab Immunol. 2003 May;10(3):411-6. doi: 10.1128/cdli.10.3.411-416.2003. PMID 12738640
- [Background] Nanan R, Rauch A, Kampgen E, Niewiesk S, Kreth HW. A novel sensitive approach for frequency analysis of measles virus-specific memory T-lymphocytes in healthy adults with a childhood history of natural measles. J Gen Virol. 2000 May;81(Pt 5):1313-9. doi: 10.1099/0022-1317-81-5-1313. PMID 10769074
- [Background] van Els CA, Nanan R. T cell responses in acute measles. Viral Immunol. 2002;15(3):435-50. doi: 10.1089/088282402760312322. PMID 12479394
- [Background] Moss WJ, Cutts F, Griffin DE. Implications of the human immunodeficiency virus epidemic for control and eradication of measles. Clin Infect Dis. 1999 Jul;29(1):106-12. doi: 10.1086/520136. PMID 10433572
- [Background] Berkelhamer S, Borock E, Elsen C, Englund J, Johnson D. Effect of highly active antiretroviral therapy on the serological response to additional measles vaccinations in human immunodeficiency virus-infected children. Clin Infect Dis. 2001 Apr 1;32(7):1090-4. doi: 10.1086/319591. Epub 2001 Mar 19. PMID 11264038
- [Background] Melvin AJ, Mohan KM. Response to immunization with measles, tetanus, and Haemophilus influenzae type b vaccines in children who have human immunodeficiency virus type 1 infection and are treated with highly active antiretroviral therapy. Pediatrics. 2003 Jun;111(6 Pt 1):e641-4. doi: 10.1542/peds.111.6.e641. PMID 12777579
- [Background] Gans H, Yasukawa L, Rinki M, DeHovitz R, Forghani B, Beeler J, Audet S, Maldonado Y, Arvin AM. Immune responses to measles and mumps vaccination of infants at 6, 9, and 12 months. J Infect Dis. 2001 Oct 1;184(7):817-26. doi: 10.1086/323346. Epub 2001 Aug 22. PMID 11528592
- [Background] Angel JB, Walpita P, Lerch RA, Sidhu MS, Masurekar M, DeLellis RA, Noble JT, Snydman DR, Udem SA. Vaccine-associated measles pneumonitis in an adult with AIDS. Ann Intern Med. 1998 Jul 15;129(2):104-6. doi: 10.7326/0003-4819-129-2-199807150-00007. No abstract available. PMID 9669968
- [Background] Moss WJ, Clements CJ, Halsey NA. Immunization of children at risk of infection with human immunodeficiency virus. Bull World Health Organ. 2003;81(1):61-70. Epub 2003 Mar 11. PMID 12640478
- See also: University of North Carolina website — http://www.unc.edu